CLINICAL TRIAL: NCT00095381
Title: A Phase II, Multi-Center Open-Label, Repeat-Dose of Forodesine Hydrochloride (BCX-1777) Infusion in Patients With Advanced T-Cell Leukemia With an Option of Long-Term Forodesine Hydrochloride (BCX-1777) Use
Brief Title: Repeat-Dose of Forodesine Hydrochloride (BCX-1777) Infusion in Patients With Advanced T-Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-T-04-201; NCT00086788 (obsolete NCT alias)
Record Dates: First submitted 2004-11-03; First posted 2004-11-04 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Leukemia, T-Cell
Keywords: Leukemia, Lymphocytic, T-Cell; Entry Term Lymphocytic Leukemia, T-Cell; T-Cell Leukemia; T-Lymphocytic Leukemia; Leukemia, Lymphocytic, T Cell; T Lymphocytic Leukemia; BCX-1777; forodesine hydrochloride; BioCryst
MeSH Terms: conditions — Leukemia, T-Cell | interventions — forodesine

INTERVENTIONS:
Drug: forodesine hydrochloride (BCX-1777)

SUMMARY:
BCX-1777 may stop the growth of cancer cells by blocking the enzymes necessary for their growth. The Phase II trial is designed to study the effectiveness of BCX-1777 in treating patients who have recurrent or refractory advanced T-cell leukemia.

Patients will receive an infusion of BCX-1777 on days 1-5. Treatment may be repeated every week for up to six courses. Patients are not required to be hospitalized for the administration of BCX-1777. Some patients may continue to receive an infusion of BCX-1777 twice a week for 6 weeks.

DETAILED DESCRIPTION:
BCX-1777 may stop the growth of cancer cells by blocking the enzymes necessary for their growth. The Phase II trial is designed to study the effectiveness of BCX-1777 in treating patients who have recurrent or refractory advanced T-cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Documented T-cell leukemia (precursor T-lymphoblastic leukemia/lymphomia or T-PLL)
* Failure to have responded to one or more standard regimens for their disease.
* Performance status of <=2 by Eastern Cooperative Oncology Group (ECOG) criteria
* All ages are eligible
* Life expectancy of at least 3 months
* Adequate liver function (aspartate transaminase [AST] and/or alanine transaminase [ALT] not >3 times upper limits or normal [ULN])
* Adequate kidney function (calculated creatinine clearance >50 mL/min)
* Negative urine pregnancy test within 2 to 7 days prior to the start of study treamtment in females of childbearing potential
* Females of childbearing potential and males must be willing and able to use an adequate method of contraception to avoid pregnancy for the duration of the study
* Signed informed consent/assent form (ICF) prior to start of any study specific procedures

Exclusion Criteria:

* Patients with known HIV infection or human T-cell leukemia virus type (HTLV-1)
* Patients with known Hepatitis B and/or Hepatitis C active infection
* Patients with active CMV infection
* Tumor-related central nervous system (CNS) leukemia requiring active treatment
* Active serious infection not controlled by oral or IV antibiotics
* Treatment with any investigational anti-leukemic agent or chemotherapy agent within 7 days prior to study entry, unless full recovery from side effects has occurred.
* Rapidly progressive disease with compromised organ function judged to be life-threatening by the investigator
* Concurrent treatment with other anticancer agents (corticosteroid use will not be excluded, but patient must remain on the stable dose)
* Cutaneous T-cell lymphoma (CTCL) diagnosis (including Sezary Syndrome)
* Pregnant and/or lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine the sustained effectiveness of IV forodesine hydrochloride infusions in patients with advanced T-cell leukemia (T-ALL or T-PLL)

SECONDARY OUTCOMES:
Safety and tolerability
Pharmacokinetics (PK) and Pharmacodynamics (PD)
maintenance of response and safety in long-term treatment

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - Los Angeles, California
  - Palo Alto, California
  - Denver, Colorado
  - Gainesville, Florida
  - Lecanto, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Rolla, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Weil Medical College of Cornell University, New York, New York
  - New York, New York
  - Syracuse, New York
  - The Bronx, New York
  - Spartanburg, South Carolina
  - Austin, Texas
  - Houston, Texas
  - Abingdon, Virginia
- Tbilisi, Georgia, Georgia